CLINICAL TRIAL: NCT00561548
Title: Impact of Anti-TNF Antibodies on the T-lymphocyte and Macrophage Cooperation in the Crohn Disease
Brief Title: Impact of Anti-Tumor Necrosis Factor (TNF) Antibodies on the T-lymphocyte and Macrophage Cooperation in Crohn Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Département de la Recherche Clinique et de l'Innovation, CHU de Nice
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 06 - PP - 2006; 2006-006877-26
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2009-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Patients with active Crohn disease and with azathioprine treatment
  Interventions: Procedure: rectosigmoïdal biopsies
- B (Other): Patient with active crohn disease and without azathioprine disease
  Interventions: Procedure: rectosigmoïdal biopsies

INTERVENTIONS:
Procedure: rectosigmoïdal biopsies — rectosigmoïdal biopsies

SUMMARY:
The aim of this research is to study Crohn disease patients before and after anti-TNF, the cooperation between lamina propria T-lymphocytes and macrophages, through the expression of co-signalisation molecules and their ligands, the production of cytokines participating in this cooperation, and the potential role of regulatory T lymphocytes.

DETAILED DESCRIPTION:
Crohn disease is an inflammatory disease and its frequency has been increasing over the last 25 years. The physiopathology involves a failure in the negative regulatory mechanisms of the inflammatory responses in the intestines, along with an excessive production of TNF-α by T-lymphocytes and macrophages of the lamina propria.

Anti-TNF-α antibodies usually give good therapeutic results, in particular in patients who are resistent or dependant on steroids. Nevertheless, in Crohn disease, the destructive T-lymphocytes - macrophage interactions, their inhibition by anti-TNFα, and the impact of these antibodies on cellular signaling remain largely unknown.

Two groups of 10 patients with active Crohn disease, with or without azathioprine, and requiring the start of anti-TNF treatment are included in this study. Rectosigmoïdal biopsies and blood tests will be done before starting the treatment and after 10 weeks of treatment. Surface antigens, cytokines and cellular molecules and the number of apoptotic cells will be analyzed by FACS, and the quantification of RNA will be analyzed by RT-PCR.

This will therefore enable us to study, before and after anti-TNF-α, in patients treated or not with azathioprine, on intestinal and blood lymphocytes, the production of cytokines involved in the lymphocyte-macrophage interaction, and the potential role of regulatory T cells.

ELIGIBILITY:
Inclusion Criteria:

* patient older than 18
* social security
* active Crohn disease defined by a CDAI > 250
* sigmoïdal and/or rectal lesions
* requiring treatment by infliximab
* having never received any anti-TNF treatment
* a negative pregnancy test for women
* prescription of efficient contraception for women, having started at least a month before beginning the study, and throughout the duration of the study
* acceptance to participate in this research and having signed the consent form
* not participating in any other study

Exclusion Criteria:

* consent withdrawal
* the halt of infliximab treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-05 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Relative variation (%) in apoptotic cells calculated according to the formula: (% of induced apoptotic cells) - (% of spontaneous apoptotic cells) | before treatment and 10 weeks after treatment

SECONDARY OUTCOMES:
Lymphocyte activation markers and macrophage activation markers | before treatment and 10 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Hébuterne, Professor, Principal Investigator — Centre Hospitalier Universitaire
Locations (1):
- Fédération des Maladies de l'appareil Digestif et de la Nutrition, Nice, France

REFERENCES:
- [Background] Puntis J, McNeish AS, Allan RN. Long term prognosis of Crohn's disease with onset in childhood and adolescence. Gut. 1984 Apr;25(4):329-36. doi: 10.1136/gut.25.4.329. PMID 6706211
- [Background] Rubin GP, Hungin AP, Kelly PJ, Ling J. Inflammatory bowel disease: epidemiology and management in an English general practice population. Aliment Pharmacol Ther. 2000 Dec;14(12):1553-9. doi: 10.1046/j.1365-2036.2000.00886.x. PMID 11121902
- [Background] Arnott ID, Watts D, Satsangi J. Azathioprine and anti-TNF alpha therapies in Crohn's disease: a review of pharmacology, clinical efficacy and safety. Pharmacol Res. 2003 Jan;47(1):1-10. doi: 10.1016/s1043-6618(02)00264-5. PMID 12526855
- [Background] ten Hove T, van Montfrans C, Peppelenbosch MP, van Deventer SJ. Infliximab treatment induces apoptosis of lamina propria T lymphocytes in Crohn's disease. Gut. 2002 Feb;50(2):206-11. doi: 10.1136/gut.50.2.206. PMID 11788561
- [Background] MacDonald TT, Di Sabatino A, Gordon JN. Immunopathogenesis of Crohn's disease. JPEN J Parenter Enteral Nutr. 2005 Jul-Aug;29(4 Suppl):S118-24; discussion S124-5, S184-8. doi: 10.1177/01486071050290S4S118. PMID 15980273
- [Background] Powrie F, Leach MW, Mauze S, Menon S, Caddle LB, Coffman RL. Inhibition of Th1 responses prevents inflammatory bowel disease in scid mice reconstituted with CD45RBhi CD4+ T cells. Immunity. 1994 Oct;1(7):553-62. doi: 10.1016/1074-7613(94)90045-0. PMID 7600284
- [Background] Noguchi M, Hiwatashi N, Liu Z, Toyota T. Secretion imbalance between tumour necrosis factor and its inhibitor in inflammatory bowel disease. Gut. 1998 Aug;43(2):203-9. doi: 10.1136/gut.43.2.203. PMID 10189845
- [Background] Itoh J, de La Motte C, Strong SA, Levine AD, Fiocchi C. Decreased Bax expression by mucosal T cells favours resistance to apoptosis in Crohn's disease. Gut. 2001 Jul;49(1):35-41. doi: 10.1136/gut.49.1.35. PMID 11413108
- [Background] Baert FJ, D'Haens GR, Peeters M, Hiele MI, Schaible TF, Shealy D, Geboes K, Rutgeerts PJ. Tumor necrosis factor alpha antibody (infliximab) therapy profoundly down-regulates the inflammation in Crohn's ileocolitis. Gastroenterology. 1999 Jan;116(1):22-8. doi: 10.1016/s0016-5085(99)70224-6. PMID 9869598
- [Background] Filippi J, Mambrini P, Arab K, Schneider SM, Hebuterne X. [Treatment of oesophageal Crohn's disease by infliximab]. Gastroenterol Clin Biol. 2005 Jan;29(1):84-5. doi: 10.1016/s0399-8320(05)80701-8. No abstract available. French. PMID 15738903
- [Background] Mitoma H, Horiuchi T, Hatta N, Tsukamoto H, Harashima S, Kikuchi Y, Otsuka J, Okamura S, Fujita S, Harada M. Infliximab induces potent anti-inflammatory responses by outside-to-inside signals through transmembrane TNF-alpha. Gastroenterology. 2005 Feb;128(2):376-92. doi: 10.1053/j.gastro.2004.11.060. PMID 15685549
- [Background] Agnholt J, Kaltoft K. Infliximab downregulates interferon-gamma production in activated gut T-lymphocytes from patients with Crohn's disease. Cytokine. 2001 Aug 21;15(4):212-22. doi: 10.1006/cyto.2001.0919. PMID 11563881
- [Background] Lugering A, Schmidt M, Lugering N, Pauels HG, Domschke W, Kucharzik T. Infliximab induces apoptosis in monocytes from patients with chronic active Crohn's disease by using a caspase-dependent pathway. Gastroenterology. 2001 Nov;121(5):1145-57. doi: 10.1053/gast.2001.28702. PMID 11677207
- [Background] Danese S, Sans M, Scaldaferri F, Sgambato A, Rutella S, Cittadini A, Pique JM, Panes J, Katz JA, Gasbarrini A, Fiocchi C. TNF-alpha blockade down-regulates the CD40/CD40L pathway in the mucosal microcirculation: a novel anti-inflammatory mechanism of infliximab in Crohn's disease. J Immunol. 2006 Feb 15;176(4):2617-24. doi: 10.4049/jimmunol.176.4.2617. PMID 16456024
- [Background] Filippi J, Roger PM, Schneider SM, Durant J, Breittmayer JP, Benzaken S, Bernard A, Dellamonica P, Hebuterne X; Groupe d'Etude Nicois Polyvalent en Infectiologie (GENPI). Infliximab and human immunodeficiency virus infection: Viral load reduction and CD4+ T-cell loss related to apoptosis. Arch Intern Med. 2006 Sep 18;166(16):1783-4. doi: 10.1001/archinte.166.16.1783. No abstract available. PMID 16983059
- [Background] Makita S, Kanai T, Oshima S, Uraushihara K, Totsuka T, Sawada T, Nakamura T, Koganei K, Fukushima T, Watanabe M. CD4+CD25bright T cells in human intestinal lamina propria as regulatory cells. J Immunol. 2004 Sep 1;173(5):3119-30. doi: 10.4049/jimmunol.173.5.3119. PMID 15322172
- [Background] Kelsen J, Agnholt J, Hoffmann HJ, Romer JL, Hvas CL, Dahlerup JF. FoxP3(+)CD4(+)CD25(+) T cells with regulatory properties can be cultured from colonic mucosa of patients with Crohn's disease. Clin Exp Immunol. 2005 Sep;141(3):549-57. doi: 10.1111/j.1365-2249.2005.02876.x. PMID 16045746
- [Background] Ochsenkuhn T, Goke B, Sackmann M. Combining infliximab with 6-mercaptopurine/azathioprine for fistula therapy in Crohn's disease. Am J Gastroenterol. 2002 Aug;97(8):2022-5. doi: 10.1111/j.1572-0241.2002.05918.x. PMID 12190171
- [Background] Rutgeerts P, Van Assche G, Vermeire S. Optimizing anti-TNF treatment in inflammatory bowel disease. Gastroenterology. 2004 May;126(6):1593-610. doi: 10.1053/j.gastro.2004.02.070. PMID 15168370